CLINICAL TRIAL: NCT03422068
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 1015550 in Patients With Idiopathic Pulmonary Fibrosis (IPF) on no Background Anti-fibrotic Therapy.
Brief Title: This Study Tests Different Doses of BI 1015550 in Patients With Idiopathic Pulmonary Fibrosis (IPF). The Study Tests How BI 1015550 is Taken up by the Body and How Well it is Tolerated.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1305-0012; 2017-002736-16 (EudraCT Number)
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18 mg BI 1015550 (Experimental): 3 tablets of 6 milligram (mg) of BI 101550 (total: 18 mg) were administrated as an oral dose together with about 240 milliliter (mL) of water twice daily (bid). Treatment period was 4 weeks for patients entered after approval of a global protocol amendment 3 at 12 Feb 2019 or 12 weeks for those entered before approval.
  Interventions: Drug: BI 1015550
- Placebo (Placebo Comparator): 3 tablets of Placebo, matching in size and weight to BI 1015550 6 milligram (mg) tablet, were administrated as an oral dose together with about 240 milliliter (mL) of water twice daily. Treatment period was 4 weeks for patients entered after approval of a global protocol amendment 3 at 12 Feb 2019 or 12 weeks for those entered before approval.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1015550 — 3 tablets of 6 milligram (mg) of BI 101550 (total: 18 mg) were administrated as an oral dose together with about 240 milliliter (mL) of water twice daily (bid).
  Other Names: Nerandomilast; JASCAYD®
  Arms: 18 mg BI 1015550
Drug: Placebo — 3 tablets of Placebo, matching in size and weight to BI 1015550 6 milligram (mg) tablet, were administrated as an oral dose together with about 240 milliliter (mL) of water twice daily.
  Arms: Placebo

SUMMARY:
The primary objective is to investigate safety and tolerability of BI 1015550 in patients with IPF.

The secondary objectives are to evaluate the pharmacokinetics (PK) of BI 1015550 in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent prior to admission to the study in accordance with ICH Harmonised Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local legislation
* Male or female patients aged ≥40 years at visit 1.
* A clinical diagnosis of IPF based on ATS/ERS/JRS/ALAT 2011 guideline within the previous 5 years as confirmed by the investigator based on chest high-resolution computed tomography (HRCT) scan taken within 12 months of visit 1 and confirmed by central review prior to visit 2.
* Forced Vital Capacity (FVC) ≥50% of predicted normal at visit 1
* Diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for haemoglobin [Hb] [Visit 1]): > 30% of predicted normal at visit 1

Exclusion Criteria:

* Patients with a significant disease or condition other than IPF which in the opinion of the investigator, may put the patient at risk because of participation, interfere with study procedures, or cause concern regarding the patient's ability to participate in the study.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Surgery of the GI tract that could interfere with PK of the trial medication (except appendectomy)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to mood disorders.
* Evidence of active infection (chronic or acute) based on clinical exam or laboratory findings.
* History of allergy or hypersensitivity to the trial medication or its excipients
* Use of drugs within 30 days prior to administration of trial medication that are known to influence the results of the trial including time between start of the Q-wave and the end of the T-wave in an electrocardiogram (QT) / QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB) (QTc)
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Participation in another trial where an investigational drug has been administered within 30 days or less than 5 half-lives (whichever is greater) of the respective drug prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug.
* Inability to refrain from smoking on trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Active drug abuse
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Inability to comply with dietary regimen required for the trial
* Patient is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male patients who do not agree to minimize the risk of female partners becoming pregnant from first dosing day until two months after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive used for at least two months prior), true sexual abstinence (when this is in line with the preferred and usual lifestyle of the patient), or surgically sterilized, including vasectomy.
* Females who are not surgically sterilised or who are not postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of Follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory).
* Relevant airways obstruction (i.e. pre-bronchodilator FEV1/FVC <0.7) at visit 1
* Patients who have previously been treated with nintedanib or pirfenidone within 30 days of visit 1.
* Positive fecal occult blood (no retest allowed),
* Positive testing for hematuria if confirmed by microscopic urine analysis (retest allowed)
* Any lifetime history of suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior)
* Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought without method, intent or plan; active suicidal thought with method, but without intent or plan; active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, intent and plan).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Odense University Hospital, Odense, Denmark
- Finland (2):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - TYKS, Turku
- Germany (2):
  - Fraunhofer ITEM, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
- Poli Univ A. Gemelli, Roma, Italy
- Netherlands (2):
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Spain
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, placebo-controlled, multiple rising dose trial was to test safety and tolerability of BI 1015550 in patients with idiopathic pulmonary fibrosis under dosage of 18mg and 24mg twice daily (bid). Dose escalation was stopped after the 18 mg bid dose group as predefined stopping criteria was met.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Participant flow was based on treatment period.
Period: Overall Study
Arm/Group | Placebo | 18 mg BI 1015550
Started | 5 | 10
Completed | 5 | 8
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Inconvenience to frequent study visits | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients who received at least one dose of study drug. It was used for the analysis of safety, demographic data, and baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 18 mg BI 1015550 | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (3.3) | 69.5 (10.1) | 69.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs) On-treatment
Description: The analysis of AEs was based on the concept of treatment-emergent AEs (TEAEs). All AEs which occurred through the treatment phase and throughout the residual effect period (REP) were considered as on treatment. Treatment period was 4 weeks for patients entered after approval of a global protocol amendment at 12 Feb 2019 or 12 weeks for those entered before approval.
Time Frame: From first dose until last dose of treatment period (duration depends on the time a patient entered the trial) + 7 days of REP or until patient's trial termination date, whichever occurred earlier, up to 35 or 91 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | 18 mg BI 1015550 | Placebo
Number analyzed (Participants) | 10 | 5
Percentage of participants | 90.0 | 60.0

2. Secondary Outcome: Area Under the Concentration-time Curve (AUCτ,1) of the BI 1015550 in Plasma Over a Uniform Dosing Interval τ After Administration of the First Dose on Day 1
Description: Area under the concentration-time curve (AUCτ,1) of the BI 1015550 in plasma over a uniform dosing interval τ after administration of the first dose on Day 1.
Time Frame: On Day 1, within 2 hours before morning dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after morning dose.
Population: Pharmacokinetic parameter set (PKS): This patient set included all patients in the TS who provided at least one pharmacokinetic (PK) parameter that was not excluded because of protocol deviations relevant to the analysis of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hours (h) / Litre (L)
Arm/Group | 18 mg BI 1015550
Number analyzed (Participants) | 10
nanomol (nmol) * hours (h) / Litre (L) | 1990 (18.2)

3. Secondary Outcome: Maximum Measured Concentration (Cmax) of the BI 1015550 in Plasma on Day 1
Description: Maximum measured concentration (Cmax) of the BI 1015550 in plasma on Day 1.
Time Frame: On Day 1, within 2 hours before morning dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after morning dose.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) / Litre (L)
Arm/Group | 18 mg BI 1015550
Number analyzed (Participants) | 10
nanomol (nmol) / Litre (L) | 277 (23.1)

4. Secondary Outcome: Area Under the Concentration-time Curve (AUCτ,ss) of the BI 1015550 in Plasma at Steady State Over a Uniform Dosing Interval τ on Day 14
Description: Area under the concentration-time curve (AUCτ,ss) of the BI 1015550 in plasma at steady state over a uniform dosing interval τ on Day 14.
Time Frame: On Day 14, within 2 hours before morning dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after morning dose.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hours (h) / Litre (L)
Arm/Group | 18 mg BI 1015550
Number analyzed (Participants) | 10
nanomol (nmol) * hours (h) / Litre (L) | 3720 (49.5)

5. Secondary Outcome: Maximum Measured Concentration (Cmax,ss) of the BI 1015550 in Plasma at Steady State Over a Uniform Dosing Interval τ on Day 14
Description: Maximum measured concentration (Cmax,ss) of the BI 1015550 in plasma at steady state over a uniform dosing interval τ on Day 14.
Time Frame: On Day 14, within 2 hours before morning dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after morning dose.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) / Litre (L)
Arm/Group | 18 mg BI 1015550
Number analyzed (Participants) | 10
nanomol (nmol) / Litre (L) | 460 (41.7)

ADVERSE EVENTS:
Time Frame: From first dose until last dose of treatment period (duration depends on the time a patient entered the trial) + 7 days of REP or until patient's trial termination date, whichever occurred earlier, up to 35 or 91 days.
Description: Treatment period was 4 weeks for patients entered after approval of the global protocol amendment 3 at 12 Feb 2019 or 12 weeks for those entered before approval. Treated set (TS): This patient set included all patients who received at least one dose of study drug. It was used for the analysis of safety, demographic data, and baseline characteristics.
Arm/Group | Placebo | 18 mg BI 1015550
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/10
Other Adverse Events (participants affected / at risk) | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | 18 mg BI 1015550 (N=10)
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | 18 mg BI 1015550 (N=10)
Bradycardia (Cardiac disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Faeces soft (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 3
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 4
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1
General physical condition decreased (Investigations) | 0 | 1
Occult blood positive (Investigations) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was halted after the first dose group (18 milligram (mg) of BI 1015550 twice daily (bid)) as the predicted gMean (based on pharmacokinetic modelling) for the next higher dosage group (24mg bid) exceeded the predefined exposure threshold.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03422068/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03422068/SAP_001.pdf